CLINICAL TRIAL: NCT00351533
Title: A Randomized, Double-blind Study of the Effect of Fish Oil (Eicosapentaenoic Acid and Docosahexanoic Acid) on Lung and Systemic Inflammation in Patients With Acute Lung Injury (ALI)
Brief Title: A Phase II Randomized Trial of Fish Oil in Patients With Acute Lung Injury (ALI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Thoracic Society (Other); Acute Respiratory Distress Syndrome Foundation (Other); American Society for Parenteral and Enteral Nutrition (Other)
Responsible Party: Principal Investigator, Renee Stapleton, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28503-A; 05-7895-A 03
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Respiratory Distress Syndrome, Adult; Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Respiratory distress syndrome, adult; Acute lung injury; Acute respiratory distress syndrome; ARDS, human; Fish oils; Fatty Acids, Omega-3; Docosahexaenoic Acids; Eicosapentaenoic Acid
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Fish Oils; Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Enteral fish oil
  Interventions: Drug: Fish oil (eicosapentaenoic acid and docosahexanoic acid)
- 2 (Placebo Comparator): Enteral saline
  Interventions: Drug: Fish oil (eicosapentaenoic acid and docosahexanoic acid)

INTERVENTIONS:
Drug: Fish oil (eicosapentaenoic acid and docosahexanoic acid) — Liquid fish oil 7.5cc enterally every 6 hours

SUMMARY:
The purpose of this study is to determine whether fish oil (containing omega-3 fatty acids) given enterally is safe and effective in reducing lung and systemic inflammation seen in acute lung injury.

DETAILED DESCRIPTION:
Acute lung injury (ALI) is common among critically ill patients and is associated with a high case fatality. Only one intervention has been shown to improve survival in a large clinical trial, and new therapies targeting the inflammatory response are needed. Nutrient interventions may provide benefit; specifically there is plausible biologic rationale for administering n-3 fatty acids (n-3 FAs) found in fish oil to patients with ALI, as n-3 FAs decrease formation of eicosanoid inflammatory mediators. However, although promising results have emerged from prior studies, fish oils have only been tested in ALI patients in a commercial enteral formula containing additional nutrients, and the control group received a high-fat enteral formula that may have been proinflammatory. Therefore, no conclusion can be drawn about the independent effect of fish oils. Furthermore, the inclusion of key pharmaconutrients in feeding formulas, instead of delivering them separately as pharmaceuticals, limits exposure to the agent, as intensive care unit (ICU) patients commonly receive less than 60% of prescribed caloric needs. Finally, specialized feeding formulas are very expensive, and it may be substantially cheaper to administer pharmaconutrients separately. We believe it is time to begin to approach nutrient trials in critically ill patients differently -- to move away from including them in feeding formulas and begin delivering them like pharmaceuticals. With appropriate scientific investigation and the use of non-nutrient placebos, this novel and innovative approach is a new paradigm of investigating nutrient delivery to critically ill patients.

This study is a phase II randomized controlled trial to determine the effects of enteral eicosapentaenoic acid (EPA) and docosahexanoic acid (DHA), both n-3 FAs found in fish oil, versus placebo on the pulmonary and systemic environments, and on clinical outcomes, in patients with ALI. We will investigate the effect of fish oil administration on several biological markers of injury and inflammation in bronchoalveolar lavage fluid and serum, on pulmonary physiologic outcomes, and on clinical outcomes.

Comparison(s): Mechanically ventilated patients with acute lung injury randomized to receive enteral fish oil versus compared to mechanically ventilated patients with acute lung injury randomized to receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Requiring positive-pressure mechanical ventilation
* ALI criteria: PaO2/FiO2 <300, bilateral infiltrates on chest radiograph, no left atrial hypertension
* Age > 17 years

Exclusion Criteria:

* Expected ICU length of stay <48 hours
* Unable to undergo bronchoalveolar lavage at enrollment
* Unable to obtain enteral access
* Post-cardiac arrest with suspected significant anoxic brain injury
* Expected survival < 28 days
* Pregnant
* Platelet count < 30,000, active bleeding, or international normalized ratio (INR)>3.0
* History of ventricular tachycardia or fibrillation
* Receiving recombinant human activated protein C (rh-APC) for sepsis
* Acquired immune deficiency syndrome (AIDS) with CD4 count < 200
* Metastatic cancer
* History of bone marrow, lung, liver, cardiac, kidney, or pancreas transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee D. Stapleton, MD, MSc, Principal Investigator — University of Vermont
Locations (5):
- United States (4):
  - St. Alphonsus Medical Center, Boise, Idaho
  - Oregon Health Sciences University, Portland, Oregon
  - University of Vermont/Fletcher Allen Health Care, Burlington, Vermont
  - Harborview Medical Center, Seattle, Washington
- St. Michael's Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Enteral Fish Oil: 7.5cc of enteral fish oil every 6 hours equalling 9.75g EPA and 6.75g DHA daily
- Enteral Saline: 7.5cc 0.9% saline every 6 hours
Period: Overall Study
Arm/Group | Enteral Fish Oil | Enteral Saline
Started | 41 | 49
Completed | 39 (Pts did not undergo BALs if not intubated) | 44 (Pts did not undergo BALs if not intubated)
Not Completed | 2 | 5
Not completed — Extubated before first BAL | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteral Fish Oil | Enteral Saline | Total
Number analyzed (Participants) | 41 | 49 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 49.0 (16.5) | 50.7 (16.5) | 49.9 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 24 | 33 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Bronchoalveolar Lavage Fluid (BALF) Interleukin (IL)-8
Description: 30 patients in the fish oil group and 36 patients in the enteral saline group underwent the 2nd bronchoalveolar lavage (BAL). Participants did not undergo BALs after baseline if they were not intubated or had expired, but clinical followup data (e.g. mortality) were collected.
Time Frame: Days 1 and 5
Population: The primary outcome was >=50% reduction in BALF IL-8, measured as the change from baseline to day 5. With α=0.05 and β=0.2, we calculated that 26 patients per group were needed if participants underwent two BALs. Analysis was intention to treat (ITT).
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | 43 [-656 to 604] | -241 [-807 to 349]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in BALF Leukotriene B4
Description: as for outcome 1
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | 6 [-1 to 14] | -2 [-26 to 9]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in BALF Interleukin-6
Description: as for outcome 1
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | -24 [-340 to 51] | -200 [-692 to 0]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in BALF Monocyte Chemotactic Protein-1
Description: as for outcome 1
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | -150 [-1812 to 93] | -226 [-752 to -38]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in BALF Neutrophil Count
Description: as for outcome 1
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: # of cells/mm^3
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
# of cells/mm^3 | -3 [-19 to 12] | -10 [-21 to 7]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Static Lung Compliance
Description: 30 patients in the fish oil group and 36 patients in the enteral saline group remained intubated on day 5 and had this outcome available.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: L/cm H20
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
L/cm H20 | 31.8 (10.1) | 36.3 (20.1)
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.26, t-test, 2 sided

7. Secondary Outcome: Oxygenation
Description: PaO2/FiO2 is the ratio of partial pressure of arterial oxygen to the fraction of inspired oxygen. 30 patients in the fish oil group and 36 patients in the enteral saline group remained intubated on day 5 and had this outcome available.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: PaO2/FiO2
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
PaO2/FiO2 | 215.4 (92.8) | 174.0 (63.4)
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

8. Secondary Outcome: Change in Plasma Interleukin-8
Description: 30 patients in the fish oil group and 36 patients in the enteral saline group underwent 2nd blood draw on day 5. Participants did not undergo blood draws after baseline if they were discharged from the ICU or had expired, but clinical followup data (e.g. mortality) were collected.
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | 0 [-8 to 0] | 0 [-13 to 0]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Plasma Leukotriene B4
Description: as for outcome 8
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | 21 [0 to 32] | -6 [-35 to 7]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Plasma Interleukin-6
Description: as for outcome 8
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | -33 [-162 to -13] | -78 [-163 to -29]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Plasma Surfactant Protein D
Description: as for outcome 8
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | 25 [0 to 32] | 36 [1 to 139]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Plasma vonWillebrand Factor
Description: as for outcome 8
Time Frame: Days 1 and 5
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 30 | 36
pg/mL | 15 [-103 to 158] | 68 [21 to 206]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Worst Multiple Organ Dysfunction Score (MODS) During First 28 Days After Study Enrollment
Description: Full scale name is Multiple Organ Dysfunction Score (MODS), a scale measuring degree of organ dysfunction in critically ill patients.
  Minimum score is 0 and maximum score is 24, with 0 indicating no organ failure and 24 indicating severe failure of multiple organs.
Time Frame: Throughout hospital stay
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 41 | 48
Scores on a scale | 8.5 (3.1) | 8.1 (3.3)
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.56, t-test, 2 sided

14. Secondary Outcome: Ventilator-free Days During First 28 Days After Study Enrollment
Description: Ventilator-free days is a common outcome measure in critical care research. A ventilator-free day is a day that a participant is alive and not receiving mechanical ventilation during the first 28 days after s/he enrolled in the study.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 41 | 48
Days | 14.5 (10.3) | 13.6 (9.9)
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.69, t-test, 2 sided

15. Secondary Outcome: ICU-free Days During First 28 Days After Study Enrollment
Description: ICU-free days is a common outcome measure in critical care research. An ICU-free day is a day that a participant is alive and not in the intensive care unit (ICU) during the first 28 days after s/he enrolled in the study.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 41 | 48
Days | 12.2 (9.8) | 11.2 (9.7)
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

16. Secondary Outcome: Hospital Length of Stay
Time Frame: At end of hospital admission
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 41 | 48
Days | 23 (18.3) | 27.6 (20.6)
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.27, t-test, 2 sided

17. Secondary Outcome: Hospital Mortality
Time Frame: At end of hospitalization
Measure: Number; unit: Participants
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 41 | 48
Participants | 9 | 10
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.65, Chi-squared

18. Secondary Outcome: 60-day Mortality
Time Frame: 60 days from day of enrollment into study
Measure: Number; unit: Participants
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 41 | 45
Participants | 9 | 11
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.49, Chi-squared

19. Secondary Outcome: Change in Bronchoalveolar Lavage Fluid (BALF) Interleukin (IL)-8
Description: 15 patients in the fish oil group and 27 patients in the enteral saline group underwent the 3rd bronchoalveolar lavage (BAL). Participants did not undergo BALs after baseline if they were not intubated or had expired, but clinical followup data (e.g. mortality) were collected.
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | -531 [-1308 to 94] | -298 [-870 to 397]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change in BALF Leukotriene B4
Description: as for outcome 19
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | 0 [-2 to 33] | 16 [0 to 50]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.38, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Change in BALF Interleukin-6
Description: as for outcome 19
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | -52 [-898 to 0] | -198 [-865 to -17]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Change in BALF Monocyte Chemotactic Protein-1
Description: as for outcome 19
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | -402 [-1690 to -41] | -670 [-1057 to -151]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Change in BALF Neutrophil Count
Description: as for outcome 19
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: # of cells/mm^3
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
# of cells/mm^3 | -4 [-48 to 8] | -10 [-56 to 15]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Change in Plasma Interleukin-8
Description: 15 patients in the fish oil group and 27 patients in the enteral saline group underwent 3rd blood draw on day 9. Participants did not undergo blood draws after baseline if they were discharged from the ICU or had expired, but clinical followup data (e.g. mortality) were collected.
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | -1 [-17 to 0] | 0 [-15 to 2]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Change in Plasma Leukotriene B4
Description: as for outcome 24
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | 10 [3 to 40] | 6 [-22 to 14]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Change in Plasma Interleukin-6
Description: as for outcome 24
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | -83 [-174 to 14] | -78 [-163 to -29]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)

27. Secondary Outcome: Change in Plasma Surfactant Protein D
Description: as for outcome 24
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | 26 [-12 to 78] | 17 [-36 to 68]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Change in Plasma vonWillebrand Factor
Description: as for outcome 24
Time Frame: Days 1 and 9
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Enteral Fish Oil | Enteral Saline
Number analyzed (Participants) | 15 | 27
pg/mL | 116 [-9 to 235] | 43 [-21 to 164]
Statistical Analysis 1: Comparison: Enteral Fish Oil vs Enteral Saline; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 28 days from day of study enrollment
Arm/Group | Enteral Fish Oil | Enteral Saline
Serious Adverse Events (participants affected / at risk) | 12/41 | 10/49
Other Adverse Events (participants affected / at risk) | 24/41 | 27/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enteral Fish Oil (N=41) | Enteral Saline (N=49)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 2 (2) | 1 (1)
Renal failure requiring renal replacement therapy (Renal and urinary disorders) | 2 (2) | 2 (2)
Pleural and pericardial effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Critical hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Trombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fulminant liver failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Right eye blindness after prolonged prone surgery (Eye disorders) | 1 (1) | 0 (0)
Recurrent falls (Nervous system disorders) | 0 (0) | 1 (1)
Aspiration with reintubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nosocomial sepsis (Infections and infestations) | 1 (1) | 1 (1)
PEA arrest (Cardiac disorders) | 1 (1) | 0 (0)
Erythema multiforme minor (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Delayed spinal cord contusion and injury (Nervous system disorders) | 1 (1) | 0 (0)
Severe hypotension (Vascular disorders) | 1 (1) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Retroperitoneal hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enteral Fish Oil (N=41) | Enteral Saline (N=49)
Total Infections (Infections and infestations) | 24 (51) | 27 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No